CLINICAL TRIAL: NCT06143969
Title: Ultrasound-assisted, Catheter-directed Thrombolysis for Acute Intermediate-high-risk Pulmonary Embolism (USAT IH-PE): Impact on Short- and Long-term Outcome, a Multi-center Experience. An Observational Retrospective and Prospective Multi-center Study
Brief Title: Ultrasound-assisted, Catheter-directed Thrombolysis for Acute Intermediate-high-risk Pulmonary Embolism
Acronym: USAT IH-PE
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 652-28112022
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; intermediate high-risk; Ultrasound-assisted; Catheter-directed Thrombolysis
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EkoSonicTM Endovascular System (EKOSTM, Boston Scientific): Patients hospitalized with acute intermediate-high risk PE treated with ultrasound-assisted, catheter-directed thrombolysis using EKOSTM.
  Interventions: Procedure: ultrasound-assisted, catheter-directed thrombolysis

INTERVENTIONS:
Procedure: ultrasound-assisted, catheter-directed thrombolysis — After 10 hours of alteplase infusion and EKOSTM ultrasound, the therapy is stopped, the EKOSTM catheter is removed, and the puncture site (internal jugular vein or femoral vein) has to be compressed.
  Other Names: EkoSonicTM Endovascular System (EKOSTM, Boston Scientific)

SUMMARY:
The purpose of this retrospective and prospective multicenter study is to evaluate the incidence of pulmonary hypertension (PH) within 6 months from ultrasound-assisted, Catheter-directed Thrombolysis for acute intermediate- high-risk Pulmonary Embolism

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) is a potentially life-threatening disease spanning a wide spectrum of clinical outcomes. PE is the third most common cardiovascular disorder in Europe and USA and causes an estimated 150,000 to 200,000 deaths.

In the latest 2019 European Society of Cardiology (ESC) Guidelines patients diagnosed with PE are stratified into different risk groups according to clinical history, hemodynamic status, cardiac biomarkers and imaging assessment of right ventricular (RV) function.

Traditionally, reperfusion therapy with systemic thrombolysis is the treatment of choice in high-risk PE, defined by sustained systemic arterial hypotension, cardiogenic shock, or the need for cardiopulmonary resuscitation.

In the setting of intermediate-risk PE,characterized by the absence of hemodynamic instability but elevated cardiac biomarkers or RV disfunction at imaging, the ESC guidelines recognize two sub-categories: intermediate-high if both signs are identified or intermediate-low, if only one of them is present.Approximately one quarter of hemodynamically stable patients with PE are at intermediate-risk, with mortality rates ranging from 3% to 15% if imaging or biomarker evidence of RV dilatation or dysfunction is present.4,5 In this subset of patients the optimal treatment strategy is still an object of debate.

A combination of ultrasound- based fragmentation of the thrombus and catheter-directed thrombolysis, requiring a reduced dose of the thrombolytic agent, has been developed. This localized therapy is currently recommended by the ESC guidelines (class IIa, LOE C) for patients with high-risk PE and contraindications for systemic thrombolysis or intermediate-high-risk PE and hemodynamic deterioration on anticoagulation treatment.

The investigators propose an observational cohort study aimed at assessing the impact on short and long-term outcome of ultrasound-assisted, catheter-directed thrombolysis using EKOSTM in a real-word population of subjects with acute intermediate-high risk PE treated in multiple Italian centers.

ELIGIBILITY:
Inclusion Criteria

* Patients admitted with acute intermediate-high risk PE, defined according to ESC guidelines
* Symptoms onset within previous 14 days associated or not with deep venous thrombosis
* Confirmation of the PE by contrast-enhanced computed tomography of the chest with embolus located in at least one main or proximal lower lobe pulmonary artery
* Echocardiographic parameters of RV disfunction
* Patients with high-risk PE or hemodynamic deterioration on anticoagulation, who have absolute contraindications (high bleeding risk) to systemic thrombolysis and symptoms onset during the last 14 days. Patients with surgery-related embolic complications are also included (within 48 hours).

Exclusion Criteria

* Age < 18 years old
* Patients unable to give informed consent
* Pregnancy
* Patients received fibrinolytic drugs in the preceding 4 days
* Bleeding diathesis
* Known bleeding disorder
* Low platelet count (< 100.000/uL
* Gastrointestinal bleeding in the preceding 3 month
* Any ongoing known presence of malignant neoplasia months
* Advanced chronic kidney disease (defined as 11.000/uL)
* Gastrointestinal bleeding in the preceding 3 month
* Any ongoing known presence of malignant neoplasia at admission with survival rate < 6
* Advanced chronic kidney disease (defined as eGFR < 30 ml/min or on dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized with intermediate high-risk pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
development of pulmonary hypertension | 6 months from treatment
  number of cases

SECONDARY OUTCOMES:
changes of echocardiographic parameters | 24 hours after the treatment and at 3-6 months follow-up
  * tricuspid annular plane excursion (TAPSE) (mm)
  * right ventricle/left ventricle ratio (RV/LV) ratio (decimal)
  * acceleration time (ACT) time (seconds)
  * fractional area change (FAC)
  * S' TDI RV (cm/sec)
  * pulmonary artery systolic pressure (PAPs) (mmHg)
  * tricuspid regurgitant velocity (TRV) (m/s)
death | within 6 months from treatment
  death during hospital stay (number of events)
death | within 6 months from treatment
  death from any cause (cancer, sepsis, respiratory failure, other) number of events
PE | within 6 months from treatment
  PE recurrence (number of events)
Major bleeding within 6 months from treatment (Bleeding Academic Research Consortium-major bleedings defined as BARC 3-5 events; clinically relevant non major bleedings defined as BARC 2 event) (number of events) | within 6 months from treatment
  Bleeding Academic Research Consortium-major bleedings defined as BARC 3-5 events; clinically relevant non major bleedings defined as BARC 2 event (number of events)
stroke | within 6 months from treatment
  number of events
Re-hospitalization | within 6 months from treatment
  Re-hospitalization (number of events)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No